CLINICAL TRIAL: NCT05944744
Title: The Role of Cobamamide Supplements in Malnourished Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Collaborators: Interbat Pharmaceuticals (Unknown)
Responsible Party: Principal Investigator, Marcellus Simadibrata, Prof. PhD., SpPD, KGEH, Professor, Fakultas Kedokteran Universitas Indonesia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-10-1267
Record Dates: First submitted 2023-02-12; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — cobamamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The patient is given Cobamamide 2 x 3000 mg for 28 days.
  Interventions: Drug: Adenosylcobalamin
- Control (Placebo Comparator): The patient is given placebo 2 x 1 capsule for 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Adenosylcobalamin — The drug contains Cobamamide / Adenosylcobalamin with dose of 3000 mg.
  Other Names: Cobazim 3000
  Arms: Intervention
Drug: Placebo — The drug doesn't contain any properties or substances for treatment.
  Arms: Control

SUMMARY:
The trial is conducted to observe the effectiveness of cobamamide supplements in improving the clinical state malnourished patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 70 years old
* Diagnosis of malnutrition based on 2019 GLIM criteria
* Participant agree to join the trial by signing infomed consent.

Exclusion Criteria:

* Malignancy (ECOG IV) and bowel obstruction
* Patients who unable to tolerate oral intake and in total parenteral nutrition
* Bowel disorder that caused severe malabsorbtion
* Patients who refuse to join the trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Change of Appetite | 28 days
  Using the Council on Nutrition Appetite Questionnaire to evaluate the appettite changes
Nutritional Status | 28 days
  Using the Subjective Global Asssessment form to assess the changes in nutritional status
Bioimpendance Analysis Result | 28 days
  Changes in Muscle Mass
Vitamin B12 (1) | 28 days
  Serum B12 Level
Vitamin B12 (2) | 28 days
  Methylmalonic Acid Level
Pre-albumin | 28 days
  Prealbumin Level
Laboratory result (1) | 28 days
  Serum ureum and creatinine level
Laboratory result (2) | 28 days
  ALT and AST level
Laboratory result (3) | 28 days
  Complete Blood Count

IPD SHARING:
Plan to Share IPD: No